CLINICAL TRIAL: NCT04528784
Title: Transcutaneous Tibial Nerve Stimulation for the Treatment of Bladder Storage Symptoms in People With Multiple Sclerosis: Protocol of a Single-arm Feasibility Study
Brief Title: Feasibility Study of Transcutaneous Tibial Nerve Stimulation for Urinary Symptoms in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Katie Robinson, Senior lecturer, Occupational therapy, University of Limerick
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTNS in MS
Record Dates: First submitted 2020-08-17; First posted 2020-08-27 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Bladder Dysfunction; Neurogenic Bladder Dysfunction; Urinary Incontinence; Urinary Bladder, Overactive; Urinary Incontinence, Urge; Nocturia; Urinary Frequency More Than Once at Night; Lower Urinary Tract Symptoms; Multiple Sclerosis; Urinary Bladder, Neurogenic
Keywords: Multiple sclerosis; Neurogenic bladder; Feasibility study; Tibial nerve stimulation
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urinary Incontinence, Urge; Nocturia; Lower Urinary Tract Symptoms; Multiple Sclerosis; Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Single-arm feasibility study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Transcutaneous tibial nerve stimulation will be applied as follows: 18 sessions of 30 minutes duration, delivered three times a week over a 6 week period using TENS device with 10 Hertz (Hz), and pulse width 200µs. The intensity of stimulation will be at the sensory and motor threshold by tingling sensation on sole of the foot with flexion of big toe and /or fanning of other toes.
  Interventions: Device: Transcutaneous tibial nerve stimulation

INTERVENTIONS:
Device: Transcutaneous tibial nerve stimulation — Transcutaneous tibial nerve stimulation is a non-invasive electrical stimulation of the posterior tibial nerve, a branch of the sciatic nerve via sacral plexus. In our study the tibial nerve will be stimulated using Transcutaneous Electrical Nerve Stimulation (TENS) unit with two surface adhesive electrodes. The anode will be positioned between 5-10 cm above medial malleolus and posterior to the edge of the tibia and the cathode will be positioned distally on arch of the foot .
  Other Names: Stimulation of tibial nerve.

SUMMARY:
Neurogenic lower urinary tract dysfunction is common among people with Multiple sclerosis with a pooled prevalence of 68.41% using self-report measures and 63.95% using urodynamic studies. Transcutaneous Tibial Nerve Stimulation (TTNS) is a non-invasive treatment option to manage bladder storage symptoms, however, the potential efficacy of TTNS among people with multiple sclerosis is based on a small number of studies with the absence of high-quality evidence relating to efficacy, and lack of clarity of the optimal electrical stimulation parameters and frequency, duration and number of treatment sessions. The feasibility and acceptability of TTNS to manage storage bladder symptoms using Transcutaneous Electrical Nerve Stimulation (TENS) needs to be established before proceeding with a definitive randomised trial. This study aims to assess whether TTNS is feasible and acceptable as a treatment for bladder storage symptoms in people with MS

DETAILED DESCRIPTION:
The investigators will use a single-arm experimental study to explore the feasibility and acceptability of TTNS in the treatment of bladder storage symptoms in multiple sclerosis. The CONSORT extension for pilot and feasibility studies will be followed to standardise the conduct and reporting of the study. The recruitment plan is twofold: 1) Open recruitment for people with MS through MS Ireland's communication channels; 2) Recruitment from a convenience sample of people with MS who have previously participated in a qualitative study. The investigators will assess recruitment/retention rates, the urinary symptoms changes and the effect on quality of life using International classification of incontinence questionnaire - overactive bladder (ICIQ-OAB), 3-day bladder diary, King's Health Questionnaire and collect self-reported data on adherence and adverse events and acceptability of using TTNS.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of any type of Multiple Sclerosis
* Male or female
* Aged ≥18 years old
* Ambulatory
* At least one bladder storage related symptom (e.g. urinary frequency, urinary urgency, nocturia with or without incontinence).

Exclusion Criteria:

* People with an indwelling urethral catheter or indwelling suprapubic catheter
* Urologic disease including bladder malignancy
* Diabetic mellitus
* Pregnant women or planning to be pregnant during the study time
* Recent pelvic related surgery <1 year
* Pacemaker or other metallic internal devices
* Urinary tract infections (UTIs) during recruitment phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Recruitment rate/ retention rate | 6 weeks
  The proportion of participants who are recruited to the study and the proportion of participants who are lost to follow up
Adherence rate | 6 weeks
  The proportion of participants who adhere to the treatment protocol of 6 weeks
Adverse events | 6 weeks
  Number of participants with adverse events as a measure of safety
Acceptability of using TTNS: proportion of participants with MS reporting that TTNS is acceptable | 6 weeks
  The proportion of participants with MS reporting that TTNS is acceptable.

SECONDARY OUTCOMES:
International Consultation of Incontinence Questionnaire-Overactive bladder (ICIQ-OAB) | 6 weeks
  Changes in the severity of scores for bladder storage symptoms experienced by participants measured using ICIQ-OAB. It has grade A for validity, reliability and responsiveness to change established with rigour on one data set. The total score ranges from 0 to 16 with higher values indicating increased symptom severity. Bother scales are not incorporated in the overall score.
Kings Health Questionnaire | 6 weeks
  Changes in scores for the effect of urinary symptoms in activity of daily living measured by the Kings Health Questionnaire. Each domain within the Kings Health Questionnaire is scored on a 0 (best) to 100 (worst) scale. A change from baseline of 5 points or higher on most of the King's Health Questionnaire domains represents a clinically meaningful improvement in health-related quality of life after treatment.
3- day bladder diary | 6 weeks
  Number of episodes of frequency, nocturia, and incontinence/ 72 hours will be calculated and compared from baseline with higher values indicating increased symptom severity.
Patient Perception of Intensity of Urgency Scale | 6 weeks
  Number of urgency episodes and severity of urgency/72 hours will be calculated and compared from baseline. The total score ranges from 0 to 4 with higher values indicating increased symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Robinson, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, LK, Ireland

REFERENCES:
- [Derived] Al Dandan HB, Galvin R, Robinson K, McClurg D, Coote S. Feasibility and acceptability of transcutaneous tibial nerve stimulation for the treatment of bladder storage symptoms among people with multiple sclerosis. Pilot Feasibility Stud. 2022 Jul 30;8(1):161. doi: 10.1186/s40814-022-01120-1. PMID 35908067
- [Derived] Al Dandan HB, Galvin R, Robinson K, McClurg D, Coote S. Transcutaneous tibial nerve stimulation for the treatment of bladder storage symptoms in people with multiple sclerosis: Protocol of a single-arm feasibility study. HRB Open Res. 2020 Sep 16;3:66. doi: 10.12688/hrbopenres.13107.1. eCollection 2020. PMID 33117961